CLINICAL TRIAL: NCT00293163
Title: A Post-Market Study to Evaluate Adverse Event Incidence Rates in Patients With Skin of Color Undergoing Correction of Nasolabial Folds With Hylaform, Hylaform Plus and Captique.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Inamed Aesthetics (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYLA00204
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Facial Wrinkles

INTERVENTIONS:
Device: Hylaform, Hylaform Plus (hylan B gel)

SUMMARY:
To assess the likelihood of keloid and scar formation, pigmentation disorders and hypersensitivity reactions in patients with skin of color undergoing correction of facial soft tissue contour deficiencies with Hylaform, Hylaform Plus or Captique.

ELIGIBILITY:
Inclusion Criteria:

* bilateral nasolabial folds with severity score 3 or 4 on the 6-point grading scale

Exclusion Criteria:

* pregnant/lactating women
* patients who previously received permanent facial implants or using over-the-counter products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
no difference in keloid and scar formation
pigmentation disorders
hypersensitivity reactions in patients with skin color compared to other patients when treated for wrinkle correction with Hylaform, Hylaform Plus or Captique

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - Grekin Skin Institute, Warren, Michigan
  - Society Hill Dermatology, Philadelphia, Pennsylvania